CLINICAL TRIAL: NCT04002323
Title: Real Life Study of Dolutegravir Plus Lamivudine in HIV-1-Infected Treatment-Naive Patients
Acronym: DOLAVI
Status: Completed | Type: Observational
Sponsor: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Carmen Hidalgo Tenorio, SPECIALIST PHYSICIAN, University Hospital Virgen de las Nieves
Other Study IDs: DOLAVI
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-1 ART-Naive: Lamivudine (300 mg p.o. q 24 h) plus Dolutegravir (50 mg p.o. q 24 h)
  Interventions: Drug: Dolutegravir 50mg Tab; Drug: Lamivudine 300 mg

INTERVENTIONS:
Drug: Dolutegravir 50mg Tab — The subjects starts their ART with this drugs, once a day
Drug: Lamivudine 300 mg — The subjects starts their ART with this drugs, once a day

SUMMARY:
Thanks to the actual highly active antiretroviral therapy (HAART) patients living with HIV have a better life expectancy, becoming chronical patients. Today's antiretroviral treatment (ART) must be maintained for life to prevent disease progression until a cure is reached. Given this need, ARTs are becoming safer and more effective but are still toxic. Cause of that simplification therapies are real, reducing the number of different Antiretrovirals involved controlling the infection. This strategies include from monotherapy using/with protease inhibitors (PI), which was investigated with treatment-experienced patients and virologically suppressed, to dual therapies which recently were investigated in treatment-naïve and treatment-experienced patients with combinations such as dolutegravir (DTG) plus lamivudine (3TC), Dolutegravir plus rilpivirine or rilpivirine plus darunavir/ritonavir boosted.

Nowadays dual therapy in real life (not into the context of a clinical trial) with dolutegravir plus lamivudine is largely studied in treatment-experienced patients who are virologically suppressed and got nearly a 100% efficacy results. Recently published results from clinical trials in treatment-naïve patients GEMINI 1 &2, where efficacy of the dual therapy with DTG 50mg plus 3TC 300mg/QD was compared versus the efficacy of triple therapy with tenofovir disoproxil fumarate, emtricitabine and dolutegravir (TDF/FTC+ DTG) (QD). Both trials show similar efficacy results, with virologic suppression higher than 90% at week 48.

Clinical trials are the gold standard to approve and add to the clinical practice new drugs and new therapies, but is also known that have some inconvenient like strict inclusion-exclusion criteria which put the study population far from being a real sample. Studies with real world data (RWD) have several strengths such as quality in medical attention and works like a bridge between clinical trials and standard clinical care, reducing/lowering general costs, improving results and accelerating the generation of knowledge.

For all the reasons above, the primary objective of this study is to analyze in treatment-naïve HIV patients the effectiveness in real life of 3TC (300 mg p.o. q 24 h) plus DTG (50 mg p.o. q 24 h). Secondary objectives are: to describe the patient who receive this dual therapy, to quantify the time gap between the clinic visit and the first dose of dual therapy administrated evaluating this dual therapy as candidate to "test and treat" therapies; to analyze the viral load drop and the increase of cluster of differentiation 4 (CD4) T lymphocytes levels; To analyze virological failures and previous mutations influence in basal resistance tests; and finally a pharmacoeconomic analysis, safety of the treatment and adherence to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (<17 y.o.)
2. Antiretroviral-naïve.
3. Be able to comply with protocol requirements and instructions.
4. Subject or the subject's representative capable of giving signed informed consent.

Exclusion Criteria:

1. Women who are breastfeeding or plan to become pregnant during the study.
2. Patients who in the investigator's judgment, poses a significant drop out risk or life expectancy inferior to study ending.
3. Patients with anticipated need to change the ART before study ending.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in approximately 139 HIV-1 infected, ART-naive adults who began their ART with DTG 50mg plus 3TC 300mg , without limits of viral load or CD4 lymphocytes recount at screening.
  The following population will be assessed:
  Intent-to-treat (ITT) Population: This population will consist of all randomized subjects who receive at least one dose of study medication.
  Intent-to-treat modified (ITT-m) Population: this population will consist of subjects in the ITT Population with the exception of mild protocol violators, those who discontinue for reasons other than those related to treatment (such as adverse events, tolerability or lack of efficacy).
  Per protocol (PP) Population: This population will consist of subjects in the ITT Population with exception of major protocol violators, such as violations which could affect the assessment of antiviral activity.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with plasma HIV 1 RNA <50 copies/milliliter at week 48 | 48 weeks
  The proportion of subjects with viral suppression (HIV-1 RNA <50 copies/mL) among subjects who received at least one dose of study medication

SECONDARY OUTCOMES:
Changes from baseline in lymphocytes cell counts at week 24 and 48 | Baseline, 24 weeks and 48 weeks
Number of Participants With Any Adverse Event (AE) | 48 weeks
  An AE is any untoward medical occurrence in a clinical investigation participant
Number of Participants Who Discontinue Treatment | 48 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Universitario Virgen de Las Nieves, Granada, Andalusia
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Clínico Universitario "Virgen de la Arrixaca", El Palmar, Murcia
  - Hospital Reina Sofía, Murcia, Murcia
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital de Jerez, Cadiz
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Campus de la Salud, Granada
  - Hospital Comarcal Santa Ana de Motril, Granada
  - Hospital de Jaen, Jaén
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Costa del Sol, Málaga
  - Hospital Comarcal de Melilla, Melilla
  - Hospital Universitario de melilla, Melilla
  - Hospital General Universitario Santa Lucía, Murcia
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Deeks SG, Lewin SR, Havlir DV. The end of AIDS: HIV infection as a chronic disease. Lancet. 2013 Nov 2;382(9903):1525-33. doi: 10.1016/S0140-6736(13)61809-7. Epub 2013 Oct 23. PMID 24152939
- [Background] Zicari S, Sessa L, Cotugno N, Ruggiero A, Morrocchi E, Concato C, Rocca S, Zangari P, Manno EC, Palma P. Immune Activation, Inflammation, and Non-AIDS Co-Morbidities in HIV-Infected Patients under Long-Term ART. Viruses. 2019 Feb 27;11(3):200. doi: 10.3390/v11030200. PMID 30818749
- [Background] Pasquau J, Hidalgo-Tenorio C. Nuke-Sparing Regimens for the Long-Term Care of HIV Infection. AIDS Rev. 2015 Oct-Dec;17(4):220-30. PMID 26679853
- [Background] Pasquau J, Hidalgo-Tenorio C, Montes ML, Romero-Palacios A, Vergas J, Sanjoaquin I, Hernandez-Quero J, Aguirrebengoa K, Orihuela F, Imaz A, Rios-Villegas MJ, Flores J, Farinas MC, Vazquez P, Galindo MJ, Garcia-Merce I, Lozano F, de Los Santos I, de Jesus SE, Garcia-Vallecillos C; QoLKAMON STUDY GROUP. High quality of life, treatment tolerability, safety and efficacy in HIV patients switching from triple therapy to lopinavir/ritonavir monotherapy: A randomized clinical trial. PLoS One. 2018 Apr 12;13(4):e0195068. doi: 10.1371/journal.pone.0195068. eCollection 2018. PMID 29649309
- [Background] Taiwo BO, Zheng L, Stefanescu A, Nyaku A, Bezins B, Wallis CL, Godfrey C, Sax PE, Acosta E, Haas D, Smith KY, Sha B, Van Dam C, Gulick RM. ACTG A5353: A Pilot Study of Dolutegravir Plus Lamivudine for Initial Treatment of Human Immunodeficiency Virus-1 (HIV-1)-infected Participants With HIV-1 RNA <500000 Copies/mL. Clin Infect Dis. 2018 May 17;66(11):1689-1697. doi: 10.1093/cid/cix1083. PMID 29253097
- [Background] Cahn P, Rolon MJ, Figueroa MI, Gun A, Patterson P, Sued O. Dolutegravir-lamivudine as initial therapy in HIV-1 infected, ARV-naive patients, 48-week results of the PADDLE (Pilot Antiretroviral Design with Dolutegravir LamivudinE) study. J Int AIDS Soc. 2017 May 9;20(1):21678. doi: 10.7448/IAS.20.01.21678. PMID 28537061
- [Background] Palacios R, Mayorga M, Gonzalez-Domenech CM, Hidalgo-Tenorio C, Galvez C, Munoz-Medina L, de la Torre J, Lozano A, Castano M, Omar M, Santos J. Safety and Efficacy of Dolutegravir Plus Rilpivirine in Treatment-Experienced HIV-Infected Patients: The DORIVIR Study. J Int Assoc Provid AIDS Care. 2018 Jan-Dec;17:2325958218760847. doi: 10.1177/2325958218760847. PMID 29529910
- [Background] Pasquau J, de Jesus SE, Arazo P, Crusells MJ, Rios MJ, Lozano F, de la Torre J, Galindo MJ, Carmena J, Santos J, Tornero C, Verdejo G, Samperiz G, Palacios Z, Hidalgo-Tenorio C; RIDAR Study Group. Effectiveness and safety of dual therapy with rilpivirine and boosted darunavir in treatment-experienced patients with advanced HIV infection: a preliminary 24 week analysis (RIDAR study). BMC Infect Dis. 2019 Feb 28;19(1):207. doi: 10.1186/s12879-019-3817-6. PMID 30819101
- [Background] Borghetti A, Lombardi F, Gagliardini R, Baldin G, Ciccullo A, Moschese D, Emiliozzi A, Belmonti S, Lamonica S, Montagnani F, Visconti E, De Luca A, Di Giambenedetto S. Efficacy and tolerability of lamivudine plus dolutegravir compared with lamivudine plus boosted PIs in HIV-1 positive individuals with virologic suppression: a retrospective study from the clinical practice. BMC Infect Dis. 2019 Jan 17;19(1):59. doi: 10.1186/s12879-018-3666-8. PMID 30654739
- [Background] Baldin G, Ciccullo A, Borghetti A, Di Giambenedetto S. Virological efficacy of dual therapy with lamivudine and dolutegravir in HIV-1-infected virologically suppressed patients: long-term data from clinical practice. J Antimicrob Chemother. 2019 May 1;74(5):1461-1463. doi: 10.1093/jac/dkz009. No abstract available. PMID 30726922
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Berger ML, Sox H, Willke RJ, Brixner DL, Eichler HG, Goettsch W, Madigan D, Makady A, Schneeweiss S, Tarricone R, Wang SV, Watkins J, Daniel Mullins C. Good practices for real-world data studies of treatment and/or comparative effectiveness: Recommendations from the joint ISPOR-ISPE Special Task Force on real-world evidence in health care decision making. Pharmacoepidemiol Drug Saf. 2017 Sep;26(9):1033-1039. doi: 10.1002/pds.4297. PMID 28913966
- [Result] Hidalgo-Tenorio C, Pasquau J, Vinuesa D, Ferra S, Terron A, SanJoaquin I, Payeras A, Martinez OJ, Lopez-Ruz MA, Omar M, de la Torre-Lima J, Lopez-Lirola A, Palomares J, Blanco JR, Montero M, Garcia-Vallecillos C. DOLAVI Real-Life Study of Dolutegravir Plus Lamivudine in Naive HIV-1 Patients (48 Weeks). Viruses. 2022 Mar 4;14(3):524. doi: 10.3390/v14030524. PMID 35336931